CLINICAL TRIAL: NCT02354807
Title: Efficacy of Pharmacological Stimulation of Brown and White Fat in Lean and Obese Young Adults
Brief Title: Efficacy of Pharmacological Stimulation of BAT and WAT in Lean and Obese Young Adults
Acronym: MiraBAT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Otto Muzik (Other)
Responsible Party: Sponsor-Investigator, Otto Muzik, Professor of Pediatrics & Radiology, Wayne State University
Organization: Wayne State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: WSU_OVPR1
Record Dates: First submitted 2015-01-22; First posted 2015-02-03 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Brown Fat
Keywords: BAT activation; quantitative PET imaging; Mirabegron effect on BAT
MeSH Terms: interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental group (Experimental): Subjects that undergo both cold exposure and one-time dose of 100mg of Mirabegron drug
  Interventions: Drug: Mirabegron; Other: Cold exposure

INTERVENTIONS:
Drug: Mirabegron — One-time dose of 100mg of Mirabegron
  Other Names: Myrbetriq
Other: Cold exposure — Exposure of subjects to cold temperature to induce non-shivering thermogenesis

SUMMARY:
To determine whether pharmacological stimulation of supraclavicular Brown Adipose Tissue (BAT or "Brown Fat") and subcutaneous White Adipose Tissue (WAT) using an FDA-approved beta3 agonist is as effective in increasing oxidative metabolism in BAT and WAT as is the exposure to cold, the investigators will assess the efficacy of an FDA approved beta3 agonist Mirabegron (trade name Myrbetriq, Astellas Pharma, Inc.) for increasing oxidative metabolism in supraclavicular BAT and subcutaneous WAT in lean and obese young adults.

The investigators anticipate that both methods to stimulate supraclavicular BAT and subcutaneous WAT will result in similar 18F-labeled fluoro-deoxyglucose (FDG) tracer uptake on positron emission tomography (PET) images as well as oxidative metabolism. This would demonstrate that pharmacological stimulation of BAT is effective and could lead to further, more detailed clinical trials in obese subjects.

DETAILED DESCRIPTION:
Obesity and diabetes have increased to epidemic proportions in the US and in many other countries. In addition, the comorbidities of these metabolic diseases, such as cardiovascular disease, cancer, osteoarthritis are placing a huge burden on the health and health care system of the United States. Finding new avenues for human therapeutics is thus a critical challenge. Brown adipose tissue (BAT or "Brown Fat") functions to dissipate stored chemical energy in the form of heat and serves to defend mammals from hypothermia and obesity.

It is now firmly established that humans have functional BAT that can be activated by mild cold stress and imaged by 18F-labeled fluoro-deoxyglucose (FDG) PET imaging. Moreover, it is now understood that there are two distinct types of brown fat cells: the "classical" brown fat (most common in supraclavicular fat depots) that form developmentally from a muscle-like myf5-positive lineage and brown fat cells that can appear in white adipose tissue (WAT) depots upon prolonged exposure to cold or beta-adrenergic signaling. These latter cells originate from a myf5-negative lineage and are referred to as beige cells. Recent data suggests that most adult humans might have both brown and beige fat cells that are inactive but could be activated via the adrenergic system. Once activated, thermogenesis in these cells could affect the body's energy balance and might be instrumental in weight management.

Although adrenergic activation using cold exposure has been shown to be highly effective in activating both brown and beige fat cells, it is difficult to implement in daily routine and there is a need for other, more practical, interventions. Mirabegron (trade name Myrbetriq, Astellas Pharma, Inc.) is a drug for the treatment of overactive bladder which was FDA approved in July of 2012. Mirabegron activates the beta3 adrenergic receptor in the detrusor muscle in the bladder, which leads to muscle relaxation and an increase in bladder capacity. There are reports of increased BAT FDG uptake following MIrabegron administration in both rodents and recently in humans. Because pharmacological stimulation of brown/beige fat cells might increase daily energy expenditure, this might represent a novel mechanism for weight management and eventually a new avenue for the treatment for obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 25 kg/m2 or BMI > 30 kg/m2
* Able to give study-specific informed consent
* Able to tolerate PET/CT imaging required by protocol, to be performed without sedation and
* Patients who are not on sedative, antidepressant, sedative antihistaminic or narcotic medications.

Exclusion Criteria:

* Subjects of reproductive potential, who are sexually active but unwilling and/or unable to use medically appropriate contraception, or women who are pregnant or breastfeeding
* Subjects with cardiac disease or hypertension
* Subjects with history of diabetes
* Subjects with severe renal impairment or subjects with moderate hepatic impairment
* Subjects with severe uncontrolled hypertension.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
SUV as a measure of glucose metabolism | 4 hours
  SUV value in supraclavicular BAT and subcutaneous WAT

SECONDARY OUTCOMES:
Blood Flow | 4 hours
  Blood Flow in supraclavicular BAT and subcutaneous WAT

CONTACTS AND LOCATIONS:
Overall Officials: Otto Muzik, Principal Investigator — Wayne State University
Locations (1):
- Children's Hospital of Michigan, Detroit, Michigan, United States

REFERENCES:
- [Result] Cypess AM, Weiner LS, Roberts-Toler C, Franquet Elia E, Kessler SH, Kahn PA, English J, Chatman K, Trauger SA, Doria A, Kolodny GM. Activation of human brown adipose tissue by a beta3-adrenergic receptor agonist. Cell Metab. 2015 Jan 6;21(1):33-8. doi: 10.1016/j.cmet.2014.12.009. PMID 25565203